CLINICAL TRIAL: NCT06184126
Title: Pilot Study to Investigate the Use of Virtual Reality Devices as an Adjunct to Usual Care for Patients With Sickle Cell Disease Experiencing Vaso-Occlusive Crises
Brief Title: Virtual Reality Devices as an Adjunct to Usual Care for Patients With Sickle Cell Disease Experiencing Vaso-Occlusive Crises
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Richard Gentry Wilkerson, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00106992
Record Dates: First submitted 2023-12-04; First posted 2023-12-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Pain Episode in Sickle Cell Disease; Acute Pain
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-blinded, randomized clinical control trial.
Masking Description: Once the participant has been enrolled in the study, they will be randomized to either the control arm or one of the experimental arms. No masking is being performed. Once randomization has occurred, participants, care providers, and the investigators will know which group the participants are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Immersive Virtual Reality (Experimental): Patient with sickle cell disease experiencing acute vaso-occlusive crisis randomized to this arm will participate in an active immersive application on the virtual reality headset with hand-held controllers. The active immersive application will allow the user to interact directly with the application and move through the virtual environment .The patient will be able to use the active immersive application on the device for a maximum of two hours.
  Interventions: Device: Virtual Reality Headset and Hand-Held Controllers
- Passive Immersive Virtual Reality (Experimental): Patient with sickle cell disease experiencing acute vaso-occlusive crisis randomized to this arm will participate in a passive immersive application on the virtual reality headset with hand-held controllers. The passive immersive application will not allow the user to interact directly with the application or move through the virtual environment .The patient will be able to use the passive immersive application on the device for a maximum of two hours.
  Interventions: Device: Virtual Reality Headset and Hand-Held Controllers
- Blindfold and Ear Plugs (Placebo Comparator): Patient with sickle cell disease experiencing acute vaso-occlusive crisis randomized to this arm will wear a blindfold and ear plugs. The patient will be able to remain blindfolded and earplugs for a maximum of two hours.
  Interventions: Other: Blindfolding and Noise Cancelling

INTERVENTIONS:
Device: Virtual Reality Headset and Hand-Held Controllers — Study Group-Virtual reality headset and hand-held controllers will be used as an adjuvant to pain management care.
  Other Names: Meta Quest 2
  Arms: Active Immersive Virtual Reality; Passive Immersive Virtual Reality
Other: Blindfolding and Noise Cancelling — Control group-Blindfold and noise cancelling headphones will be a placebo comparator group to the experimental interventions of virtual reality devices.
  Arms: Blindfold and Ear Plugs

SUMMARY:
This study aims to evaluate the use of virtual reality as an adjunct to standard care for patients with sickle cell disease experiencing vaso-occlusive crises.

DETAILED DESCRIPTION:
A prospective, non-blinded, non-randomized trial will be conducted at the Adult Emergency Department at the University of Maryland Medical Center and Adult Urgent Care Center, which is managed by the Department of Emergency Medicine, located in Baltimore, Maryland.

Patients meeting eligibility criteria and who have signed the research informed consent will be enrolled in this study. Subject data collected will include demographic information, symptoms of the current illness and physical exam findings.

Upon enrollment into the study, a study team member will interview the patient to collect data needed to complete the Case Report Form. Patients assigned to one of the two virtual reality study groups will be directed by research coordinators who can help with equipment as needed throughout the session. The virtual reality device will be limited to a maximum of 2 hours of use. Assessments will be made at 4 different timepoints: 1) Immediately before the intervention, 2) at the 1-hour mark of the intervention, 3) immediately after the intervention, and 4) 1 hour after the intervention. During these assessments, patients will rate their pain intensity using a 0-10 numerical scale. Additionally, at each assessment, patients will be asked to state the change in pain that has taken place since the last measurement. This measurement will be performed without informing the patient of their previously recorded pain scores.

Data will also be recorded regarding the patient's 1) comfort of the device, 2) disposition (discharged home vs observation/admission status), 3) total length of treatment time in the ED (measured as time to initiation of any treatment to the time of final disposition), and 4) total amount of opioids administered while under the care of the emergency department clinicians, converted into morphine milligram equivalents. Each patient will complete a questionnaire at the conclusion of the session regarding their perceived impact of the intervention, ease of use, and likelihood to reuse the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age > 18 years) emergency department patient
* History of sickle cell disease
* Presenting to the emergency department due to acute pain related to sickle cell disease thought to be due to vaso-occlusive crisis

Exclusion Criteria:

* Prior enrollment in this study
* Presenting with a chief complaint suggestive of a complicated crisis (such as concern for acute chest syndrome, splenic sequestration, hepatic sequestration, pulmonary embolism) as determined by the clinical care provider
* Not being treated with intravenous opioids for the vaso-occlusive crisis
* Patients who lack the capacity to provide informed consent
* Medical history of seizures or known intolerance to virtual reality
* Disabilities like vision and hearing defects etc. that preclude the use of a head mounted virtual reality device.
* Known to be pregnant
* Incarcerated at the time of evaluation
* Over the age of 89 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the change in pain scores between the 3 groups at one hour after completion of the study intervention. | A single time point 1 hour after the study intervention ends.
  Patient reported on 0-10 scale

SECONDARY OUTCOMES:
Comparison of the subject's assessment of comfort of the study intervention between the 3 groups | Immediately before intervention, at 1-hour mark of the intervention, immediately following the intervention, and 1 hour after the intervention ends.
  Patient reported on 1-5 Likert scale
Comparison of the proportion of subjects within each group who are hospitalized. | Day of enrollment
  Determine whether the patient is discharged home vs. placed in observation/admission status after completion of emergency department care.
Compare the total duration of Emergency Department treatment measured from the time of delivery of the first intervention to the time of disposition. | Day of enrollment
  Measured in hours/minutes
Comparison of the quantity opioids, converted to morphine milligram equivalents, administered while under the care of the ED clinical team. | Day of enrollment
  Measured in morphine milligram equivalents
Comparison of the change in pain scores between the 3 groups at one hour after study intervention begins. | A single time point 1 hour after the study intervention begins.
  Patient reported on 0-10 scale
Comparison of the change in pain scores between the 3 groups at completion of the study intervention. | A single time point at the completion of the study intervention.
  Patient reported on 0-10 scale

CONTACTS AND LOCATIONS:
Overall Officials: R. Gentry Wilklerson, MD, Principal Investigator — U of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Systems, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing any individual participant data with other researchers

REFERENCES:
- [Background] Sundd P, Gladwin MT, Novelli EM. Pathophysiology of Sickle Cell Disease. Annu Rev Pathol. 2019 Jan 24;14:263-292. doi: 10.1146/annurev-pathmechdis-012418-012838. Epub 2018 Oct 17. PMID 30332562
- [Background] Jang T, Poplawska M, Cimpeanu E, Mo G, Dutta D, Lim SH. Vaso-occlusive crisis in sickle cell disease: a vicious cycle of secondary events. J Transl Med. 2021 Sep 20;19(1):397. doi: 10.1186/s12967-021-03074-z. PMID 34544432
- [Background] Duroseau Y, Beenhouwer D, Broder MS, Brown B, Brown T, Gibbs SN, Jackson K, Liang S, Malloy M, Romney ML, Shani D, Simon J, Yermilov I. Developing an emergency department order set to treat acute pain in sickle cell disease. J Am Coll Emerg Physicians Open. 2021 Aug 7;2(4):e12487. doi: 10.1002/emp2.12487. eCollection 2021 Aug. PMID 34401866
- [Background] Osunkwo I, Manwani D, Kanter J. Current and novel therapies for the prevention of vaso-occlusive crisis in sickle cell disease. Ther Adv Hematol. 2020 Sep 29;11:2040620720955000. doi: 10.1177/2040620720955000. eCollection 2020. PMID 33062233
- [Background] Williams H, Tanabe P. Sickle Cell Disease: A Review of Nonpharmacological Approaches for Pain. J Pain Symptom Manage. 2016 Feb;51(2):163-77. doi: 10.1016/j.jpainsymman.2015.10.017. Epub 2015 Nov 17. PMID 26596876
- [Background] Chuan A, Zhou JJ, Hou RM, Stevens CJ, Bogdanovych A. Virtual reality for acute and chronic pain management in adult patients: a narrative review. Anaesthesia. 2021 May;76(5):695-704. doi: 10.1111/anae.15202. Epub 2020 Jul 27. PMID 32720308
- [Background] Smith V, Warty RR, Sursas JA, Payne O, Nair A, Krishnan S, da Silva Costa F, Wallace EM, Vollenhoven B. The Effectiveness of Virtual Reality in Managing Acute Pain and Anxiety for Medical Inpatients: Systematic Review. J Med Internet Res. 2020 Nov 2;22(11):e17980. doi: 10.2196/17980. PMID 33136055
- [Background] Agrawal AK, Robertson S, Litwin L, Tringale E, Treadwell M, Hoppe C, Marsh A. Virtual reality as complementary pain therapy in hospitalized patients with sickle cell disease. Pediatr Blood Cancer. 2019 Feb;66(2):e27525. doi: 10.1002/pbc.27525. Epub 2018 Oct 26. PMID 30362236
- [Background] Mercado SH. An outpatient pain plan and ED pain pathway for adults with sickle cell disease. JAAPA. 2023 Mar 1;36(3):20-23. doi: 10.1097/01.JAA.0000920956.33631.26. PMID 36752670